CLINICAL TRIAL: NCT01096433
Title: Association of Circadian Variations,Sleep Architecture, Hypertension, and Prostaglandin in Sleep Apnea
Brief Title: Circadian Variations of Prostaglandin in Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyoto University (Other)
Responsible Party: Principal Investigator, Yuichi Chihara, Medical doctor, Kyoto University
Organization: Kyoto University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-411
Record Dates: First submitted 2010-03-29; First posted 2010-03-31 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Sleep Apnea; Continuous Positive Airway Pressure; Prostaglandins; Circadian Variations
Keywords: Sleep apnea; CPAP; Prostaglandins; Circadian variations
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPAP (Experimental): The subjects introduced with CPAP treatment
  Interventions: Device: CPAP treatment

INTERVENTIONS:
Device: CPAP treatment — maintains upper airway patency and minimizes the obstructive events
  Other Names: REMstar (Respironics), Auto Set(Resmed), Goodnight (Tyco Healthcare)

SUMMARY:
The purpose of this study is to evaluate the associations of circadian variations, sleep architecture, hypertension and prostanoids in the patients with sleep apnea. In addition, the patients introduced to continuous positive airway pressure(CPAP) treatment, the effects of CPAP are also evaluated.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by repetitive episodes of upper airway obstruction during sleep that provoke frequents arousals, sleep fragmentation, oxygen desaturation, and excessive daytime sleepiness. OSA may contribute to the development of systemic hypertension, cardiovascular disease. Many studies has reported a crucial role for the prostaglandin D system in sleep regulation. In addition, it has been described urinary or blood levels of prostaglandins was higher in the patients with hypertension, diabetes mellitus, and these values were associated with the severity of coronary artery disease. However, the relation between alterations of prostaglandin D system and sleep architecture, sleepiness, and clinical outcomes such as hypertension, arteriosclerosis in the patients with OSA are not known. Additionally, after CPAP treatment, we will investigate the association between change of prostaglandin system and sleep architecture, sleepiness, clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects on admission for sleep study under the Respiratory Care and Sleep Control Medicine, Kyoto University Hospital.
* Subjects diagnosed with OSA (apnea hypopnea index >=5/hour) by overnight polysomnography.

Exclusion Criteria:

* Subjects treating for acute infections or malignancy.
* Subjects with severe cardiovascular disease, diabetes,and renal failure.
* Subjects taking nonsteroidal anti-inflammatory drugs, steroids or immunosuppressants.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Prostaglandins in the urine and blood | baseline, and 2days, 3 months after CPAP

SECONDARY OUTCOMES:
polysomnography measurements | baseline, and 2days, 3 months after CPAP
sleepiness and health-related quality of life | baseline, and 2days, 3 months after CPAP
Clinical measurements (blood pressure, heart rate, sympathetic activity etc) | baseline, and 2days, 3 months after CPAP
serum and urinary biomarker (inflammation, oxidative stress etc.) | baseline, and 2days, 3 months after CPAP
endothelial function | baseline, and 2days, 3 months after CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Chin, MD,PhD, Principal Investigator — Kyoto University, Graduate School of Medicine; Yuichi Chihara, MD, Principal Investigator — Kyoto University Hospital
Locations (1):
- Kyoto University Graduate School of Medicine, Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Chihara Y, Chin K, Aritake K, Harada Y, Toyama Y, Murase K, Yoshimura C, Hitomi T, Oga T, Mishima M, Urade Y. A urine biomarker for severe obstructive sleep apnoea patients: lipocalin-type prostaglandin D synthase. Eur Respir J. 2013 Dec;42(6):1563-74. doi: 10.1183/09031936.00133512. Epub 2012 Dec 6. PMID 23222881